CLINICAL TRIAL: NCT04152915
Title: A Trial to Demonstrate Bioequivalence Between Semaglutide D Formulations for the DV3396 Pen-Injector and the Formulation for the PDS290 Semaglutide Pen-Injector
Brief Title: A Research Study Looking at Similarity Between Once-weekly Semaglutide Versions for Different Injection Pens
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-4588; U1111-1235-3506 (Other: World Health Organization (WHO)); 2019-002588-92 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2019-11-04; First posted 2019-11-05 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteers; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DV3396 (Experimental): Semaglutide administered with the DV3396 pen-injector (semaglutide D, test formulation)
  Interventions: Drug: Semaglutide
- PDS290 (Experimental): Semaglutide administered with the PDS290 pen-injector (semaglutide reference formulation)
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Increasing doses of semaglutide administered s.c. (subcutaneouly, under the skin) once weekly for 7 weeks

SUMMARY:
The study will look at how two different semaglutide versions reach and stay in the blood after injection. The study aims to show similar levels of semaglutide in the blood when using the different semaglutide versions. Participants will get 1 of the 2 versions of semaglutide. Which version participants get is decided by chance. One version is the one that doctors already can prescribe and the other is the new version. Participants will get the medicines as an injection under the skin of the stomach with the use of a pen-injector. The type of pen-injector is different for the two versions of semaglutide. The study will last for about 80-99 days. Participants will have 24 study visits with the study doctor. For 2 of the visits, participants will stay in the clinic for 4 days and 3 nights. Participants may have to stop the study if the study doctor thinks that there are risks for their health. Women cannot take part if pregnant, breast-feeding or planning to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65 years (both inclusive) at the time of signing informed consent.
* Body mass index between 25.0 and 34.9 kg/m^2 (both inclusive) and
* Body weight between 65.0 and 130.0 kg (both inclusive).
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using highly effective contraceptive methods.
* Any disorder which in the investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol.
* Use of prescription medicinal products or non-prescription drugs, except routine vitamins, topical medications, highly effective contraceptives and occasional use of paracetamol and acetylsalicylic acid (the two latter are not allowed within 24 hours before screening), within 14 days prior to the day of screening.
* Abuse or intake of alcohol, defined as any of the below:
* Known or suspected alcohol abuse within 1 year prior to the day of screening (defined as regular intake of more than an average intake of 24 g alcohol daily for men and 12 g alcohol daily for women)
* Positive alcohol test at screening
* Abuse or intake of drugs, defined as any of the below:
* Known or suspected drug/chemical substance abuse within 1 year prior to the day of screening
* Positive drug of abuse test at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
AUC0-last,sema,1mg: Area under the semaglutide concentration time curve from time 0 until last quantifiable measurement after one dose of s.c. semaglutide 1 mg administration following a 6-week dose escalation period | 0-840 hours after one dose of s.c. semaglutide 1 mg
  hours*nmol/L
Cmax,sema,1mg: Maximum observed semaglutide concentration after one dose of s.c. semaglutide 1 mg administration following a 6-week dose escalation period | 0-840 hours after one dose of s.c. semaglutide 1 mg
  nmol/L

SECONDARY OUTCOMES:
AUC0-168h,sema,0.25mg,SS: Area under the semaglutide concentration time curve from time 0 until 168 hours at steady state after the last dose of s.c. semaglutide 0.25 mg administration | 0-168 hours after the last dose of s.c. semaglutide 0.25 mg
  hours*nmol/L
Cmax,sema,0.25mg,SS: Maximum observed semaglutide concentration at steady state after the last dose of s.c. semaglutide 0.25 mg administration | 0-168 hours after the last dose of s.c. semaglutide 0.25 mg
  nmol/L
AUC0-∞,sema,1mg: Area under the semaglutide concentration time curve from time 0 until infinity after one dose of s.c. semaglutide 1 mg administration following a 6-week dose escalation period | 0-840 hours after one dose of s.c. semaglutide 1 mg
  hours*nmol/L
tmax,sema,1mg: Time of maximum observed semaglutide concentration after one dose of s.c. semaglutide 1 mg administration following a 6-week dose escalation period | 0-840 hours after one dose of s.c. semaglutide 1 mg
  hours
tmax,sema,0.25mg,SS: Time of maximum observed semaglutide concentration at steady state after the last dose of s.c. semaglutide 0.25 mg administration | 0-168 hours after the last dose of s.c. semaglutide 0.25 mg
  hours
t½,sema,1mg: terminal elimination half-life of semaglutide after one dose of s.c. semaglutide 1 mg administration following a 6-week dose escalation period | 0-840 hours after one dose of s.c. semaglutide 1 mg
  hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Mainz, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com